CLINICAL TRIAL: NCT02847091
Title: Post-marketing Clinical Study of Ipragliflozin; Multicenter, Open-label Study to Assess the Efficacy of Ipragliflozin Add-on in Reducing Insulin Dose in Patients With Type 2 Diabetes Mellitus Receiving Insulin Therapy
Brief Title: Study of Ipragliflozin in Patients With Type 2 Diabetes Mellitus Receiving Insulin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1941-MA-3054
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Ipragliflozin; SGLT2 inhibitor; Type 2 diabetes mellitus; ASP1941
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipragliflozin Group (Experimental): Ipragliflozin will be administered orally for 24 weeks.
  Interventions: Drug: Ipragliflozin; Drug: Insulin

INTERVENTIONS:
Drug: Ipragliflozin — Oral administration, 50mg once daily
  Other Names: ASP1941; Suglat
Drug: Insulin — Patients are receiving insulin therapy from at least 12 weeks before Visit 1 (is allowed ±10% dose modification if clinically needed, and is reduced within a 20% to 40% range at Visit 1 and then is controlled up to Visit 8 based on criteria of this study).

SUMMARY:
The objective of this study is to assess the reduction in insulin dose from baseline at Week 24 while keeping the blood glucose levels controlled (maintaining HbA1c values) when ipragliflozin is administered once daily for 24 weeks in patients with type 2 diabetes mellitus receiving insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* The subject has been receiving insulin therapy for the treatment of diabetes mellitus.
* The subject has type 2 diabetes mellitus and has been receiving insulin monotherapy or insulin therapy in combination with one or two oral hypoglycemic agents.
* The subject has not modified diet or exercise therapies or dosage regimen of oral hypoglycemic agents, or has not switched to another pharmacotherapy for 12 weeks before Visit 1.
* The subject has an HbA1c value between 6.5% and <8.0%.
* The subject has a body mass index (BMI) of >23.0 kg/m2.
* If the subject is a female, she must satisfy the following criteria. The subject is not of childbearing potential and satisfies any of the following criteria.

  * The subject is post-menopausal (absence of menses for at least 1 year).
  * The subject is surgically sterile.

The subject is of childbearing potential but satisfies all of the following criteria:

* The subject agrees not to get pregnant to 28 days after the last dose of the study drug.
* The subject has a negative pregnancy test. The subject agrees to use two of the established contraceptive methods listed below to 28 days after the last dose of the study drug when having heterosexual intercourse.

  * If the subject is a female, she must agree not to breastfeed to 28 days after the last dose of the study drug.
  * If the subject is a female, she must agree not to donate their eggs during the period from the assessment to 28 days after the last dose of the study drug.
  * In case a male subject's spouse or partner is of childbearing potential, the subject must agree to use two of the established contraceptive methods to 28 days after the last dose of the study drug.
  * If the subject is a male, he must agree not to donate their sperm to 28 days after the last dose of the study drug.

Exclusion Criteria:

* The subject has type 1 diabetes mellitus.
* The subject has any symptom of dysuria, anuria, oliguria or urinary retention.
* The subject has proliferative retinopathy.
* The subject has diabetic ketoacidosis.
* The subject has a history or complication of medically significant renal disease such as renovascular occlusive disease, nephrectomy and/or renal transplant.
* The subject has a history of recurrent urinary tract infection.
* The subject has symptomatic urinary tract infection or symptomatic genital infection.
* The subject has chronic disease(s) that require the continuous use of corticosteroids, immunosuppressants, etc.
* The subject has a history of cerebral vascular attack, unstable angina, myocardial infarction, vascular intervention, and serious heart disease within 1 year (52 weeks) before signing of the informed consent.
* The subject has a complication or surgical history of serious gastrointestinal disorder.
* The subject has severe hepatic dysfunction.
* The subject has uncontrolled blood pressure.
* The subject has unstable psychiatric disorder.
* The subject has severe infection or serious trauma, or perioperative.
* The subject has drug addiction or alcohol abuse.
* The subject has a history of malignant tumors.
* The subject has a history of an allergy to ipragliflozin and/or similar drugs (drugs possessing SGLT2 inhibitory action).
* The subject has used SGLT2 inhibitors, GLP-1 receptor agonists, sulfonylureas (SU), glinide agents, or insulin products other than long-acting insulin within 12 weeks before signing of the informed consent.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin dose | Baseline and Week 24
Percent change from baseline in insulin dose | Baseline and Week 24

SECONDARY OUTCOMES:
Change from baseline in insulin dose | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20 and the last assessment during the treatment period (up to Week 24)
Percent change from baseline in insulin dose | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20 and the last assessment during the treatment period (up to Week 24)
Change from baseline in HbA1c | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in fasting plasma glucose | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in cholesterol | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in glycoalbumin | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in leptin | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in adiponectin | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in glucagon | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in C-peptide | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in body weight | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in waist circumference | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in blood pressure | Baseline and Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and the last assessment during the treatment period (up to Week 24)
Change from baseline in DTSQ | Baseline and Week 24 and the last assessment during the treatment period (up to Week 24)
  DTSQ: Diabetes treatment satisfaction questionnaire
Number of subjects achieving withdrawal of insulin therapy | Up to Week 24
Percent of subjects achieving withdrawal of insulin therapy | Up to Week 24
Safety assessed by incidence of Adverse events | Up to Week 24
Safety assessed by blood pressure in a sitting position | Up to Week 24
Safety assessed by pulse rate in a sitting position | Up to Week 24
Safety assessed by Hematology | Up to Week 24
Safety assessed by biochemistry | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (15):
- Japan (15):
  - Site JP00007, Gunma
  - Site JP00008, Hiroshima
  - Site JP00009, Hyōgo
  - Site JP00010, Kanagawa
  - Site JP00003, Mie
  - Site JP00004, Osaka
  - Site JP00015, Shiga
  - Site JP00002, Tochigi
  - Site JP00005, Tochigi
  - Site JP00013, Tochigi
  - Site JP00001, Tokyo
  - Site JP00006, Tokyo
  - Site JP00011, Tokyo
  - Site JP00012, Tokyo
  - Site JP00014, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Ishihara H, Yamaguchi S, Sugitani T, Kosakai Y. Open-Label Study to Assess the Efficacy of Ipragliflozin for Reducing Insulin Dose in Patients with Type 2 Diabetes Mellitus Receiving Insulin Therapy. Clin Drug Investig. 2019 Dec;39(12):1213-1221. doi: 10.1007/s40261-019-00851-z. PMID 31552641
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=281